CLINICAL TRIAL: NCT00057343
Title: A Prospectively Randomized, Phase III, Multicenter, Controlled Trial to Evaluate the Safety and Efficacy of the Zevalin Therapeutic Regimen Plus Rituxan Compared With Rituxan Alone in Patients With Relapsed or Refractory Follicular NHL
Brief Title: Safety and Efficacy of Zevalin in the Treatment of Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 106-10
Record Dates: First submitted 2003-03-31; First posted 2003-04-01 (Estimated); Last update posted 2006-09-12 (Estimated); Status verified 2006-09

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ibritumomab tiuxetan; Rituximab

INTERVENTIONS:
Drug: Zevalin (ibritumomab tiuxetan)
Drug: Rituxan (rituximab)

SUMMARY:
The purpose of this study is to provide treatment for patients who have relapsed NHL or refractory NHL, and to determine the effectiveness and safety of the Zevalin and Rituxan regimens or Rituxan therapy alone on your disease.

ELIGIBILITY:
Summary of major inclusion and exclusion criteria. Other Safety criteria will need to be met.

Inclusion Criteria:

* Histologically confirmed, relapsed or refractory CD20+ follicular B-cell NHL within 12 months of Study Day 1 (without clinical evidence of transformation). NHL must require treatment as determined by an increase in overall tumor size. The presence of B symptoms, and/or the presence of masses which are causing ongoing clinical symptoms.
* Bidimensionally measurable disease meeting the minimum requirement of at least 1 lesion >/= 2.0 cm in a single dimension.
* No lymphoma therapy for 3 weeks prior to Study Day 1.
* Patients must be recovered from all toxicities associated with prior surgery, radiation therapy, chemotherapy, or immunotherapy.
* Signed IRB-approved informed consent.
* Greater than 18 years of age.
* Expected survival >/= 3 months.
* WHO performance status of </= 2.
* Acceptable hematologic status, liver function, renal function, and pulmonary function.
* Female patients who are not pregnant or lactating.
* Men and women of reproductive potential who are following accepted birth control methods.

Exclusion Criteria:

* Patients with impaired bone marrow reserve, which may be indicated by prior myeloablative therapy with autologous bone marrow transplantation (ABMT) or peripheral blood stem cell (PBSC) rescue.
* Prior radioimmunotherapy, including the Zevalin regimen.
* Prior immunotherapy, including Rituxan therapy within 6 months of Study Day 1.
* Rituxan-refractory (no response to most recent Rituxan-containing regimen, or TTP was < 6 months).
* Presence of CNS lymphoma.
* Patients with chronic lymphocytic leukemia (CLL).
* Known history of HIV or AIDS.
* Serious nonmalignant disease or infection
* Major surgery, other than diagnostic surgery, within 4 weeks of Study Day 1.
* Patients who received investigational product within 4 weeks of Study Day 1 or patients who may experience long-term toxicity from a previous investigational therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2003-03

PRIMARY OUTCOMES:
Event-free survival

SECONDARY OUTCOMES:
overall response rate
complete response rate
unconfirmed complete response rate
partial response rate
duration of response
time to progression
time-to-next anticancer therapy
quality of life
overall survival
safety profile

CONTACTS AND LOCATIONS:
Locations (67):
- United States (67):
  - Research Site, Huntsville, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Bakersfield, California
  - Research Site, Concord, California
  - Research Site, Duarte, California
  - Research Site, Loma Linda, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Newport Beach, California
  - Research Site, Orange, California
  - Research Site, Sacramento, California
  - Biogen Idec Incorporated, San Diego, California
  - Research Site, San Diego, California
  - Research Site, Santa Barbara, California
  - Research Site, Vallejo, California
  - Research Site, Farmington, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Jacksonville, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Boise, Idaho
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Aurora, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Harvey, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Urbana, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Saint Joseph, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Albuquerque, New Mexico
  - Research Site, Farmington, New Mexico
  - Research Site, Buffalo, New York
  - Research Site, Manhasset, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Bismarck, North Dakota
  - Research Site, Cleveland, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Temple, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Bremerton, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Wausau, Wisconsin